CLINICAL TRIAL: NCT06623682
Title: Efficacy, Cost-effectiveness and Implementation of an Integrated Self-help and Support Services for Student Mental Health in Tertiary Institutions: JCTH+ Pragmatic Cluster RCT
Brief Title: Study of Self-Help and Support Services for Student Mental Health in Tertiary Institutions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Winnie W.S. MAK, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SBRE-23-0966A
Record Dates: First submitted 2024-09-20; First posted 2024-10-02 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Mental Health; Mental Well-being; Psychological Intervention; Self-care
Keywords: Online Psychological Intervention; Mental Health; Mental Well-being; Self-care
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- JCTH+-integrated mental health services (Experimental): In the intervention arm, the JCTH+ platform will be integrated into the existing services of tertiary education institutions and introduced to students through mass advertisement within the institution. After randomization, three tertiary education institutions are allocated in this arm, including Chinese University of Hong Kong (CUHK), University of Hong Kong (HKU), and Hong Kong University's School of Professional and Continuing Education (HKU SPACE). Students will be invited to join this study and give consent adhering to the declaration of Helsinki.
  Interventions: Behavioral: Transdiagnostic cognitive behavioural therapy
- Service-as-usual (SAU) (No Intervention): In the no-intervention group, participants will continue with their usual practice, i.e. service-as-usual (SAU), for 4 months before implementing the project. After randomization, three tertiary education institutions are allocated in this arm, including The Hong Kong Polytechnic University (PolyU), Tung Wah College (TWC) and City University of Hong Kong (CityU). The same integration procedure will be implemented after this waiting period.

INTERVENTIONS:
Behavioral: Transdiagnostic cognitive behavioural therapy — Transdiagnostic cognitive behavioural therapy for both depression and anxiety that including modules from (1) Mindfulness-based intervention, (2) Rumination-focused cognitive behavioural therapy, and also including modules for insomnia and from Mindwork (Internet-based cognitive behavioural therapy).
  Arms: JCTH+-integrated mental health services

SUMMARY:
This proposed study aims to evaluate the implementation of integrating the existing services in tertiary education institutions with the JCTH+ platform. The study aims to evaluate the efficacy of JCTH+ on students' mental health outcomes as compared to service as usual, and to assess the cost-utility of the platform to determine whether the benefits of implementing the platform justify the costs associated. It is hypothesized that participants who receive integrated self-help and support services will show (H1) a greater reduction in mental health symptoms, and (H2) better mental well-being compared with participants in the control condition, i.e. service-as-usual (SAU).

DETAILED DESCRIPTION:
This study is a parallel pragmatic cluster-randomized control trial evaluating the efficacy and cost-utility of a JCTH+-integrated services, as compared to service-as-usual among tertiary education institutions in Hong Kong. Randomisation will be carried out at institution level based on a computer-generated sequence. The estimated sample size will be 1,684, with 842 participants per condition. A factorial design will be adopted with all eligible participants completing assessments at 7 timepoints: baseline, 4 months post-test, 8-, 12-, 16-, 20- and 24-months follow-up. The primary endpoint is 4 months at post-test after baseline assessment. Concurrently, all staff involved in the project will be interviewed qualitatively at 12 months and 24 months from enrolment to understand their experience in the integration process and effectiveness of implementation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or above
* Able to read Chinese or English
* With internet connection and able to access the internet
* With moderate-severe GAD-7 a/o moderate-severe PHQ-9
* studying full-time at a tertiary education institution in Hong Kong

Exclusion Criteria:

* not able to read and understand Chinese;
* under 18 years old;
* not able to access the Internet or use digital devices
* without depressive symptoms or anxiety symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1684 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2026-08-29 (Estimated); Study Completion 2026-08-29 (Estimated)

PRIMARY OUTCOMES:
Recovery Quality of Life-20 | Baseline, 4 months, 8 months, 12 months, 16 months, 20 months and 24 months
  It measures the quality of life in individuals with mental health conditions using a 5-point scale from 0 (none of the time) to 4 (most or all of the time). It focuses on aspects crucial to those recovering from mental illness, such as well-being, self-perception, relationships, and activity. Total scores ranged from 0 to 80, where higher scores indicated higher overall quality of life. The scale is validated for its reliability and sensitivity in the Chinese-Hong Kong population, making it an effective tool for both clinical settings and research to track recovery progress and treatment outcomes in mental health in the local context.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder Assessment | Baseline, 4 months, 8 months, 12 months, 16 months, 20 months and 24 months
  It is a 7-item scale to assess the extent to which respondents are bothered by anxiety-related symptoms using a 4-point scale from 0 (not at all) to 3 (nearly every day). Scores of 5, 10, and 15 denote the mild, moderate, and severe levels of anxiety respectively (range: 0-21). At a cut-off of 10, GAD-7 has sensitivity of 0.89 and specificity of 0.82 in detecting generalized anxiety disorder (GAD). The internal consistency of the Chinese version was 0.93.
Patient Health Questionnaire | Baseline, 4 months, 8 months, 12 months, 16 months, 20 months and 24 months
  It includes 9 items to assess the extent to which respondents are bothered by depression-related symptoms using a 4-point scale from 0 (not at all) to 3 (nearly every day). PHQ-9 has been validated and used widely in the general population for screening and measuring depression severity. Scores of 5, 10, 15, and 20 denote mild, moderate, moderately severe, and severe levels of depression respectively (range: 0-27). PHQ-9 has sensitivity of 0.88 and specificity of 0.88 in detecting major depressive disorder (MDD) at a cut-off of 10. The internal consistency reliability of the Chinese version of the scale was 0.86.
Self-Stigma Of Seeking Help | Baseline, 4 months, 8 months, 12 months, 16 months, 20 months and 24 months
  It assesses the person's perception and reaction to seeking professional help using a 5-point scale from 1 (Strongly Disagree) to 5 (Strongly Agree). The SSOH consists of 10 items. Total scores ranged from 10 to 50, where higher scores indicate higher levels of self-stigma of seeking help. The measurement demonstrated good reliability and validity in previous studies.
Youth Empowerment Scale-Mental Health | Baseline, 4 months, 8 months, 12 months, 16 months, 20 months and 24 months
  The individual level subscale was adopted, which contains 6 items to assess the level of self-empowerment in mental health using a 5-point scale from 0 (Never or almost never) to 5 (Always or almost always). Total scores ranged from 6 to 30, where higher scores indicated higher level of ability in managing emotion and mental health. The scale has demonstrated good internal consistency and construct validity.
5-level EQ-5D version | Baseline, 4 months, 8 months, 12 months, 16 months, 20 months and 24 months
  The EQ-5D-5L comprises five dimensions, MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN /DISCOMFORT and ANXIETY/ DEPRESSION, each dimension has five response levels: no problems, slight problems, moderate problems, severe problems, unable to/extreme problems. The respondent is asked to indicate his/her health state by checking the box next to the most appropriate response level for each of the five dimensions. Responses are coded as single-digit numbers expressing the severity level selected in each dimension. The digits for the five dimensions can be combined in a 5-digit code that describes the respondent's health state; for instance, 21111 means slight problems in the mobility dimension and no problems in any of the other dimensions.
Nonattachment Scale-Short Form | Baseline, 4 months, 8 months, 12 months, 16 months, 20 months and 24 months
  Nonattachment Scale-Short Form (NAS-SF) includes 8 items to measure nonattachment using a 6-point Likert scale from 1 (strongly disagree) to 6 (strongly agree). Total scores ranged from 8 to 48, where higher scores indicated higher levels of nonattachment. It yielded satisfactory internal consistency and validity.
General Mattering Scale | Baseline, 4 months, 8 months, 12 months, 16 months, 20 months and 24 months
  The 5-item General Mattering Scale measures perceptions and feelings of being important to other people (e.g., "How much would you be missed if you went away?"). Items are rated on a scale ranging from 1 (Not at all) to 4 (A lot) with good reliability and validity. Total scores ranged from 5 to 20, where higher scores indicated higher level of mattering.
Anti-Mattering Scale | Baseline, 4 months, 8 months, 12 months, 16 months, 20 months and 24 months
  The Anti-Mattering Scale is a five-item scale ranging from 1 (Not at all) to 4 (A lot) assessing the degree to which people feel like they do not matter to others. Sample item include "To what extent have you been made to feel like you are invisible?". Total scores ranged from 5 to 20, where higher scores indicated lower levels of mattering.
Perceived Competence | Baseline, 4 months, 8 months, 12 months, 16 months, 20 months and 24 months
  It contains 4 items on a 7-point Likert scale from 1 (none at all) to 7 (very true) to assess the self-perceived competence in maintaining regular self-care. Total scores ranged from 4 to 28, where higher scores indicated higher levels of self-perceived competence in maintaining regular self-care.
Treatment Self-regulation Questionnaire | Baseline, 4 months, 8 months, 12 months, 16 months, 20 months and 24 months
  It contains 15 items on a 7-point Likert scale from 1 (not true at all) to 5 (completely true) to understand the reason for beginning or keeping regular mental self-care. Higher scores in each item indicate higher importance of the reason for keeping mental self-care.
Mindful Self-Care Scale | Baseline, 4 months, 8 months, 12 months, 16 months, 20 months and 24 months
  The scale utilizes a 6-point Likert scale, ranging from 0 = never to 4 = regularly, to measure self-care in six factors: physical care, supportive relationships, mindful awareness, self-compassion and purpose, mindful relaxation, and supportive structure. A higher score indicates a higher frequency of engaging in mindful self-care within the past week. The scale demonstrates adequate reliability with Cronbach's coefficient alphas equal to 0.89 for the total 33-item.
College Self-Efficacy Inventory | Baseline, 4 months, 8 months, 12 months, 16 months, 20 months and 24 months
  It evaluates the self-efficacy of college students in academic settings. It consisted of 20 items that load into three subscales: Course Efficacy, Social Efficacy, and Roommate Efficacy. In this study, only 16 items on Course Efficacy, Social Efficacy will be included since dormitory is not usually available for students at post-secondary institutions. The confidence level is measured by using a scale ranging from 1 (Not confident at all) to 10 (Extremely confident). Higher scores in each subscale demonstrate a higher level of self-efficacy in that dimension.
Basic Psychological Need Satisfaction in General | Baseline, 4 months, 8 months, 12 months, 16 months, 20 months and 24 months
  It contains 21 items to measure basic psychological need satisfaction in 3 subscales: Autonomy, Competence, and Relatedness. The scale used a 7-point Likert scale from 1 (not at all true ) to 7 (very true). Higher scores in each subscale indicated a higher degree to which the person experiences satisfaction with each of the three needs.

CONTACTS AND LOCATIONS:
Locations (1):
- Diversity and Well-being Lab, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No